CLINICAL TRIAL: NCT00911924
Title: A Prospective, Unmasked Evaluation of the iStent in Patients With Primary Open-Angle Glaucoma
Acronym: SY
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Glaukos Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Synergy; Synergy Trial
Record Dates: First submitted 2009-06-01; First posted 2009-06-03 (Estimated); Last update posted 2015-05-20 (Estimated); Status verified 2015-05

CONDITIONS: Glaucoma; Eye Diseases; Glaucoma, Open-Angle
Keywords: primary open angle glaucoma (POAG); OAG; glaucoma
MeSH Terms: conditions — Glaucoma; Eye Diseases; Glaucoma, Open-Angle | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- iStent (Experimental)
  Interventions: Device: iStent

INTERVENTIONS:
Device: iStent — Glaukos iStent, medication
  Other Names: stent, trabecular micro-bypass stent

SUMMARY:
Prospective, unmasked, evaluation of the iStent in patients that have primary open-angle glaucoma (OAG). Stent implantation in one eye will be used for analysis, with medication added at 6 months, as required.

DETAILED DESCRIPTION:
One hundred patients will be enrolled in the study at up to 21 sites; follow-up is through 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of primary open-angle glaucoma
* Male or female at least 18 years of age and able to provide written informed consent
* Mean IOP (at baseline visit after washout of any medications) must be at least 22 mm Hg and no greater than 38 mm Hg
* Likely to be available and willing to attend follow-up visits

Exclusion Criteria:

* Angle closure glaucoma
* Secondary glaucomas
* Prior glaucoma procedures
* Elevated episcleral venous pressure from history of active thyroid orbitopathy, carotid-cavernous fistula, orbital tumors, or orbital congestive disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2009-05; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
IOP 18 mm Hg or less without medications | At 6 months
IOP 18 mm Hg or less with or without medications | 12 months

SECONDARY OUTCOMES:
Mean IOP | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Jeff Wells, PharmD, MBA, Study Director — Glaukos Corporation
Locations (13):
- S.V. Malayan's Ophtalmology Centre, Yerevan, Armenia
- Allgemeines Krankenhaus Wien, Vienna, Austria
- France (3):
  - Chu de Lyon Hospital Edouard Herriot, Lyon
  - CHNO des Quinze-Vingts, Paris
  - Hopital Saint-Joseph, Paris
- Germany (4):
  - Knapschaftskrankenhaus Bochum Langendreer, Bochum
  - Universitatsklinkum Erlangen, Erlangen
  - Universitatsklinikum Magdeburg A.o.R., Magdeburg
  - Dietrich-Bonhoeffer-Klinikum Neubrandenburg, Neubrandenburg
- Italy (2):
  - Universita' degli Studi di Parma, Parma
  - Universita'di Torino, Torino
- Spain (2):
  - Hospital clinico San Carlos, Madrid
  - Hospital Torrevieja Salud, UTE, Torrevieja

REFERENCES:
- [Result] Voskanyan L, Garcia-Feijoo J, Belda JI, Fea A, Junemann A, Baudouin C; Synergy Study Group. Prospective, unmasked evaluation of the iStent(R) inject system for open-angle glaucoma: synergy trial. Adv Ther. 2014 Feb;31(2):189-201. doi: 10.1007/s12325-014-0095-y. Epub 2014 Jan 23. PMID 24452726